CLINICAL TRIAL: NCT00566189
Title: New Frontiers on Bariatric Surgical Procedures. Classical Bypass for Type 2 Diabetic Patients With BMI Between 30 and 34.9 kg/m2
Brief Title: New Frontiers on Bariatric Surgical Procedures: Classical Bypass for Type-2 Diabetic Patients With Obesity Grade I
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Campinas, Brazil (Other)
Collaborators: Ethicon Endo-Surgery (Industry)
Responsible Party: Principal Investigator, Bruno Geloneze, Prof Dr Bruno Geloneze, MD, PhD, University of Campinas, Brazil
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LIMED0004
Record Dates: First submitted 2007-11-30; First posted 2007-12-03 (Estimated); Last update posted 2013-03-08 (Estimated); Status verified 2013-03

CONDITIONS: Diabetes Mellitus, Type 2; Insulin Resistance; Obesity
Keywords: diabetes mellitus, type 2; Insulin resistance; Intra-Abdominal Fat; Omentum; duodenal exclusion; bariatric surgery; Glucagon-Like Peptide 1; Gastric Inhibitory Polypeptide; insulin; glucagon; ghrelin; adiponectin; Cytokines
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Insulin Resistance; Obesity | interventions — Gastric Bypass

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): Roux-en-Y bypass gastroplasty
  Interventions: Procedure: Roux-en-Y Bypass Gastroplasty

INTERVENTIONS:
Procedure: Roux-en-Y Bypass Gastroplasty — Under open laparotomy, a stomach section separates a 80-ml proximal gastric pouch. A jejunum section below Treitz's Angle creates an excluded gastrobiliopancreatic limb of 150cm. A Roux-in-Y retrocolic anastomosis of the alimentary limb promotes the continuity between the gastric pouch and the jejunum and a silastic ring reduces the pouch outlet.The anastomosis of the excluded limb is done 100cm below the silastic ring.
  Other Names: Roux-en-Y Gastric Bypass

SUMMARY:
Bariatric surgery leads to remission of type 2 diabetes in morbid obese patients in 80% (Roux-en-Y gastric bypass)to 90% (biliopancreatic diversion and duodenal switch) of cases. The current consensus supports bariatric surgical treatment for diabetic patients with BMI as low as 35kg/m2 but it has questioned that lower body mass patients might benefit of the surgery as well.

This study is proposed to describe the effects of Roux-en-Y gastric bypass in mild obese (BMI 30-35) human volunteers on incretins, insulin production and sensitivity and its clinical (diabetic chronic complications) and metabolic impact.

DETAILED DESCRIPTION:
Bariatric surgery leads to remission of type 2 diabetes in morbid obese patients in 80% (Roux-en-Y gastric bypass)to 90% (biliopancreatic diversion and duodenal switch) of cases; most of the remainder achieve better glycemic control, even if they regain weight. The current consensus supports bariatric surgical treatment for diabetic patients with BMI as low as 35kg/m2 but it has questioned that lower body mass patients might benefit of the surgery as well.

Actually, many clinical researchers worldwide would consider a lower limit BMI of 30kg/m2, i.e., any grade of obesity.

This study is proposed to describe the effects of Roux-en-Y gastric bypass (Fobi-Capella technique, adapted to create a larger gastric pouch, about 80ml)in mild obese (BMI 30-35) human volunteers on incretins, insulin production and sensitivity and its clinical (diabetic chronic complications) and metabolic impact.

ELIGIBILITY:
Inclusion Criteria:

* Obesity grade I (BMI 30-34,9)
* Weight variance less than 5% in the last 3 months.
* Previous diagnosis of diabetes type 2.
* Insulin requirement, alone or along with oral agents
* Capacity to understand the procedures of the study.
* To agree voluntarily to participate of the study, signing an informed consent.

Exclusion Criteria:

* Positive Anti-GAD antibodies
* Laboratorial signal of probable failure of insulin production, i. e., seric peptide C lesser than 1 ng/mL.
* History of hepatic disease like cirrhosis or chronic active hepatitis.
* Kidney dysfunction (creatinine > 1,4 mg/dl in women and > 1,5 mg/dl in men).
* Hepatic dysfunction: aspartate aminotransferase or alanine aminotransferase 3x above upper normal limit.
* Recent history of neoplasia (< 5 years).
* Use of oral or injectable corticosteroids for more than consecutive 14 days in the last three months.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2007-08; Primary Completion 2011-08 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Improvement or reversal of type 2 diabetes mellitus | 7 days, 14 days, 21 days, 1 month, 2 months, 3 months, six months and one year.

SECONDARY OUTCOMES:
Changes in body weight and fat distribution after intervention | 1 month, 2 months, 3 months, 6 months and 1 year
Changes in the secretion pattern of incretins, insulin and glucagon after intervention, as measured by standardized mixed meal tolerance test | 6 months and 1 year
Improvement of insulin sensitivity as measured by insulin tolerance test | 1 month, 3 months, 6 months and 1 year
Changes in seric free fatty acids, lipoproteins, adiponectin and other adipokines | one month, 2 months, 3 months, 6 months and 1 year
Regression of carotid intima-media thickness | 1 month, 3 months, 6 months and 1 year
Retardation of progression of disturbances of peripheral nerves as detected by electroneuromyography | 1 year and 2 years
Retardation of progression of diabetic retinal complications as detected by fundoscopy and retinography | 1 year and 2 years
Retardation of progression or regression of albuminuria as detected by microalbuminuria assay in 24-h urine collection | 6 months, 1 year and 2 years

CONTACTS AND LOCATIONS:
Overall Officials: José Carlos Pareja, MD, PhD, Principal Investigator — University of Campinas (UNICAMP); Bruno Geloneze, MD, PhD, Principal Investigator — University of Campinas (UNICAMP)
Locations (1):
- LIMED (Laboratory of Investigation of Metabolism and Diabetes)/GASTROCENTRO/Univeristy of Campinas (UNICAMP), Campinas, São Paulo, Brazil

REFERENCES:
- [Background] Pories WJ. Diabetes: the evolution of a new paradigm. Ann Surg. 2004 Jan;239(1):12-3. doi: 10.1097/01.sla.0000102990.47956.98. PMID 14685094
- [Background] Pories WJ, Swanson MS, MacDonald KG, Long SB, Morris PG, Brown BM, Barakat HA, deRamon RA, Israel G, Dolezal JM, et al. Who would have thought it? An operation proves to be the most effective therapy for adult-onset diabetes mellitus. Ann Surg. 1995 Sep;222(3):339-50; discussion 350-2. doi: 10.1097/00000658-199509000-00011. PMID 7677463
- [Background] Pories WJ, MacDonald KG Jr, Flickinger EG, Dohm GL, Sinha MK, Barakat HA, May HJ, Khazanie P, Swanson MS, Morgan E, et al. Is type II diabetes mellitus (NIDDM) a surgical disease? Ann Surg. 1992 Jun;215(6):633-42; discussion 643. doi: 10.1097/00000658-199206000-00010. PMID 1632685
- [Background] Geloneze B, Tambascia MA, Pilla VF, Geloneze SR, Repetto EM, Pareja JC. Ghrelin: a gut-brain hormone: effect of gastric bypass surgery. Obes Surg. 2003 Feb;13(1):17-22. doi: 10.1381/096089203321136539. PMID 12630608
- [Background] Geloneze B, Tambascia MA, Pareja JC, Repetto EM, Magna LA. The insulin tolerance test in morbidly obese patients undergoing bariatric surgery. Obes Res. 2001 Dec;9(12):763-9. doi: 10.1038/oby.2001.105. PMID 11743060
- [Derived] Fellici AC, Lambert G, Lima MM, Pareja JC, Rodovalho S, Chaim EA, Geloneze B. Surgical treatment of type 2 diabetes in subjects with mild obesity: mechanisms underlying metabolic improvements. Obes Surg. 2015 Jan;25(1):36-44. doi: 10.1007/s11695-014-1377-9. PMID 25098565